CLINICAL TRIAL: NCT02163343
Title: Serum Metal Ion Levels in Patients Who Underwent Cathcart/Corail Hemiarthroplasty for Fractured Neck of Femur
Status: Suspended | Type: Observational
Sponsor: Royal Berkshire NHS Foundation Trust (Other Government)
Collaborators: DePuy International (Industry)
Responsible Party: Sponsor
Other Study IDs: 14/WS/0060
Record Dates: First submitted 2014-06-06; First posted 2014-06-13 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Fractured Neck of Femur
Keywords: Serum metal ion levels; Cathcart/Corail hemiarthroplasty; Hip replacement
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
Elevated serum metal ions are well recognized in metal-on-metal articulations in total hip replacements. The objective of the study is to see if the Cathcart / Corail device implanted during a hemiarthroplasty (replacement of one half of the hip joint) results in elevated serum metal ion levels (cobalt & chromium) and to see if there is an association between size of Cathcart head used and metal ion levels.

DETAILED DESCRIPTION:
Hip hemiarthroplasty is a very common operation. The investigator's organisation (RBH) performs approximately 140 Cathcart Hemiarthroplasty procedures each year and over 500 Cathcart/Corail have been implanted since their introduction to the department in March 2010. The clinical outcome is good with a low mortality rate at both 30 days and one year. The implant is well established in the department and there has been a reduction in the need for revision procedures compared with the previously used cemented Exeter Trauma Stem (ETS).

Elevated serum metal ion levels (cobalt and chromium) are well recognised in metal-on-metal (MoM) articulations in total hip arthroplasty. The Medicines and Healthcare Products Regulatory Agency have issued guidelines on follow up of all patients who underwent either MoM total hip replacement or resurfacing. All patients must undergo serum metal ion levels testing with recommended upper limits of 119 nmol/L for cobalt and 134.5 nmol/L for Chromium. Above those levels further surveillance or revision is required. It is not known whether the large diameter Cathcart head on the Corail stem also results in elevated serum metal ion levels (above the MHRA guidelines). Research published in 2012 has demonstrated that there is excessive wear and corrosion between the trunnion and taper of the ASR XL head, which is similar in design to the Cathcart head, utilising a taper insert within the head. Concern has therefore been raised that there may be excessive wear, and increased serum metal ion levels, in patients who have undergone Cathcart hemiarthroplasty.

The investigators propose to measure serum cobalt and chromium metal ions (normal levels are under 30nmol/l) in participants who have received a Cathcart Hemiarthroplasty greater than one year ago and ask each participant to complete the twelve question Oxford hip score .This is to identify whether the levels are elevated and whether clinical scores are able to detect those patients who may have a problem related to increased metal ion levels, and to obtain a normal distribution. It is known that metal ion levels are elevated at one year and the increase can be maintained for several years subsequently following metal-on-metal total hip replacements.

From a statistical perspective, this is a pragmatic study to see if there is an association between Cathcart Hemiarthroplasty and raised serum metal ion levels.

The procedure will involve writing to the patient to invite them to enter the study. If they are interested (through return of the reply slip or telephone call from the patient to the orthopaedic office) an appointment at the hospital will be arranged. Non return of the reply slip or no telephone contact from the patient will be regarded as the patient not wishing to take part. In clinic they will be assessed and further clarity given or any questions answered before informed consent is sought. Once consent has been obtained, the patient will complete the Oxford Hip Score questionnaire and a blood test for metal ion levels will be taken.

In year 2, a letter will be sent to General Practitioner (GP) requesting whether they would be able to perform a blood test for the study. At this time the patient's status would also be established. If the GP is willing to do the blood test a reminder letter will be sent to the patient inviting them to go to the GP or hospital for the second blood test. If the GP is unable to do the blood test, the letter to the patient will only give the option of going to the hospital for the blood test.

As the investigators have a large cohort of patients it may also be possible to identify an association between head diameter, clinical outcome and the risk of having elevated metal ion levels. This is important as smaller resurfacing components (diameter less than 51 mm) are at increased risk of elevated metal ion levels and the majority of fractured neck of femur patients are female who often require small components.

* Primary outcome: Serum Cobalt and Chromium Levels at one and two years.
* Secondary outcomes: Whether there is an association between i) Oxford Hip Score at one year, and, ii) head diameter and metal ion levels.

ELIGIBILITY:
Inclusion Criteria:

* All patients who received a Cathcart Hemiarthroplasty and are able to attend for blood testing and complete a questionnaire (Oxford Hip Score).

Exclusion Criteria:

* Those patients too frail or who now live too far away to attend for blood testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients receiving a Cathcart Hemiarthroplasty for intracapsular fractured neck of femur at the Royal Berkshire Hospital
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in serum metal ion level (Chromium and Cobalt) at year 2 | One and two years post surgery

SECONDARY OUTCOMES:
The association between Oxford Hip Score, head diameter and metal ion levels. | up to two years post surgery
  Whether there is an association between i) Oxford Hip Score at one year, and, ii) head diameter and metal ion levels and year one and year two.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Andrade, FRCS MSc, Principal Investigator — Royal Berkshire NHS Foundation Trust
Locations (1):
- Royal Berkshire NHS Foundation Trust, Reading, Berkshire, United Kingdom